CLINICAL TRIAL: NCT06741527
Title: Post Market Confirmatory Interventional Clinical Study of the Integrity Implant System Used for Rotator Cuff Tear Augmentation
Brief Title: Integrity Implant System Post Market Clinical Follow-Up Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 24-01
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tears of the Shoulder
Keywords: Rotator Cuff Repair; Shoulder repair; Integrity Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Integrity Implant System (Other)
  Interventions: Device: Integrity Implant System

INTERVENTIONS:
Device: Integrity Implant System — Integrity Implant System used for Rotator Cuff Repair

SUMMARY:
The study design is a prospective, multi-center, single-arm, non-randomized post market clinical follow-up study to confirm the performance, safety and clinical benefit of the Integrity Implant System when used for rotator cuff tear augmentation (with or without repair).

DETAILED DESCRIPTION:
The Study Objective is to confirm the performance, safety and clinical benefit of the Integrity Implant System when used for rotator cuff tear augmentation (with or without repair).

The clinical success will be evaluated by absence of rotator cuff re-tear. Performance and clinical benefits will be evaluated by functional outcomes measured using standard scoring systems such as the American Shoulder and Elbow Surgeons Shoulder Score (ASES), Constant-Murley Score (CMS), Patient Satisfaction, EQ-5D-5L, Single Assessment Numeric Evaluation (SANE), Visual Analogue Scale (VAS) and rotator cuff repair outcomes measured using MRI evaluation for repair integrity, quality, tendon tissue thickness and regeneration.

Safety of the Integrity Implant System will be assessed by monitoring the frequency and incidence of adverse events.

The Primary Endpoint shall confirm the Performance of the Integrity Implant System when used for rotator cuff augmentation (with or without repair). Performance will be evaluated by an adequately powered analysis of retear rates seen by MRI at 12-months after surgery.

ELIGIBILITY:
1. At least 18 years of age
2. Able (with assistance from LAR, if necessary) to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures.
3. Able to complete all Patient Reported Outcome Measure (PROM) questionnaires.
4. Fully understands study requirements and able to return for all required follow-up visits and assessments.
5. Able to comply with all post-operative physician prescribed rehabilitation instructions.
6. Index shoulder rotator cuff tendon tear surgical access may be performed using mini-open, single-portal arthroscopic or multi-portal arthroscopic intervention
7. Meets all intended use and indications for use defined within the Integrity Implant System IFUs as applied to rotator cuff tendon tears. These include:

Index shoulder rotator cuff tendon tear needs management and protection from injury

Index shoulder has no substantial loss of tendon tissue

Index shoulder rotator cuff tendon tear footprint allows approximation of soft tissue and fixation of the Integrity Implant to tendon tissue using an Integrity Tissue Tack

Index shoulder rotator cuff tendon tear footprint allows fixation of the Integrity Implant to bone using the Integrity Bone Staple

Exclusion Criteria

The subject exclusion criteria are as follows:

1. Medical condition that in the PI's opinion would place the subject at risk or interfere with the study
2. Vulnerable population (prisoners, minors, pregnant women, mentally ill persons and the elderly or any person under any undue pressure from others to participate in the study)
3. Pregnant, breastfeeding, or plans to become pregnant during the study
4. History of poor compliance with medical treatment of any kind
5. Deemed contraindicated for MRI by the PI
6. Previous rotator cuff surgery (any type) on the index shoulder
7. Current instability of the index shoulder
8. Rotator cuff tendon tear is a Massive Cofield Classified Full-Thickness Tear (tear length >5cm)
9. Chondromalacia of index shoulder ≥ Grade 3
10. Fatty infiltration of the index shoulder rotator cuff muscle ≥ Grade 3
11. Insulin dependent Type I Diabetes
12. History of heavy smoking (≥ 1 pack per day) within last 6-months
13. History of auto-immune or immunodeficiency disorders
14. Currently taking immunosuppression medication for other diseases (e.g., transplants or other inflammatory diseases)
15. Oral steroid use in the last 2-months or injectable steroid use in the last 3-months
16. History of cognitive or mental health status that interferes with study participation
17. Poor comprehension of English language
18. Meets one or more of the contraindications defined within the Integrity Implant System IFUs as applied to rotator cuff tendon tears. These include:

18.1 Rotator cuff tendon tear is deemed irreparable by the PI

18.2 Rotator cuff tendon tear repair requires replacement of damaged tendon

18.3 Rotator cuff tendon tear repair requires fixation of soft tissue to adjoining soft tissue

18.4 Rotator cuff tendon tear repair requires tendon strength reinforcement

18.5 Presence of infection

18.6 Any condition which would limit the ability or willingness to restrict activities or follow directions during the healing period

18.7 Hypersensitivity to any of the Integrity Implant System components

18.8 Inadequate soft tissue support for Integrity Tissue Tack fixation

18.9 Inadequate quality of bone for Integrity Bone Staple fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Re-tear rate after rotator cuff augmentation | 12 months postoperatively
  Assessed by MRI evaluation at 12 months post-operatively defined using Sugaya classification system.

SECONDARY OUTCOMES:
The American Shoulder and Elbow Surgeons (ASES) Score | Screening/Pre-Op, 6 weeks, 6-month, 12-month and 24-month Post-operatively
  The American Shoulder and Elbow Surgeon's (ASES) Score is a tool used to measure shoulder function. The ASES score is on a scale of 0 to 100, with 0 being the worst possible score and 100 the best. The score consists of two components - pain and activities of daily living.
Constant-Murley Score (CMS) | Screening/Pre-Op, 6 weeks, 6-month, 12-month and 24-month post-operatively
  The Constant-Murley Shoulder Score is a scoring method used by clinicians to assess function of the shoulder. The standard score is on a scale of 0 to 100, with 0 being no shoulder function and 100 being excellent function.
EQ-5D-5L (EuroQol) | Screening/Pre-Op, 6 weeks, 6-month, 12-month and 24-month post-operatively
  The 5-level EQ-5D (EQ-5D-5L) is a standardized self-assessed, health related quality of life questionnaire. It is composed of five questions with Likert scale response options (descriptive system) and a visual analog scale (EQ-VAS). The EQ-VAS asks patients to rate their own health from 0 to 100 (the worst and best imaginable health, respectively).
The Single Assessment Numeric Evaluation (SANE) Score | Screening/Pre-Op, 6 weeks, 6-month, 12-month and 24-month post-operatively
  The Single Assessment Numeric Evaluation (SANE) Score is a tool used to assess the subject's perception of their affected joint. Participants are requested to rate their shoulder function on a scale of 0 to 100, with 0 as the worst option and 100 being normal shoulder function.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Central Indiana Orthopaedics, Fishers, Indiana
  - Towson Orthopaedic Associates/University of Maryland St. Joseph's Medical Center, Towson, Maryland
  - Virtua Health, Marlton, New Jersey
  - Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina
  - Campbell Clinic, Germantown, Tennessee